CLINICAL TRIAL: NCT05679908
Title: A Phase 2, Double-blind, Randomized, Multicenter, Placebo-controlled, Three Arm Parallel Study to Evaluate the Efficacy and Safety of TNX-1900 (Intranasal Oxytocin) in Patients With Chronic Migraine (PREVENTION Study)
Brief Title: A Study to Evaluate the Efficacy and Safety of TNX-1900 in Patients With Chronic Migraine
Acronym: PREVENTION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Collaborators: Premier (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TNX-OX-CM201
Record Dates: First submitted 2022-12-19; First posted 2023-01-11 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Chronic Migraine; Chronic Migraine, Headache; Chronic Migraine Without Aura; Aura Migraine
Keywords: Migraine; Chronic Migraine; Headache; Chronic Migraine Without Aura; Aura Migraine
MeSH Terms: conditions — Headache; Migraine with Aura; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TNX-1900 High Dose (Experimental): 30 IU oxytocin taken intranasally twice daily.
  Interventions: Drug: TNX-1900
- TNX-1900 Low Dose (Experimental): 30 IU oxytocin taken intranasally once daily. Placebo taken intranasally once daily.
  Interventions: Drug: TNX-1900; Drug: Placebo Nasal Spray
- Placebo (Placebo Comparator): Placebo taken intranasally twice daily.
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: TNX-1900 — Patients will spray TNX-1900 once into each nostril.
  Other Names: intranasal oxytocin
  Arms: TNX-1900 High Dose; TNX-1900 Low Dose
Drug: Placebo Nasal Spray — Patients will spray placebo nasal spray once into each nostril.
  Arms: Placebo; TNX-1900 Low Dose

SUMMARY:
This is a phase 2, double-blind, randomized, multicenter, placebo-controlled, three arm parallel study to evaluate the efficacy and safety of two different dosages (30 IU daily and 60 IU daily) of TNX-1900 in patients with chronic migraine.

ELIGIBILITY:
Major Inclusion Criteria:

* Men and women aged 18 to 65 years, inclusive, at the time of Visit 1.
* History of migraine with or without aura for at least 1 year and onset at < 50 years of age. Patient must also have a history of chronic migraine > 3 months prior to Visit 1 as defined by IHS ICHD-3
* Patients can be on stable ≤ 1 preventive medication and any number of abortive migraine medications for 90 days prior to Screening and during the study. All treatments, other than the study drug, thought to have preventive efficacy in migraine should not be started or discontinued during the entire study period. Note: Up to approximately 30% of the patients randomized into the study can be on 1 preventative medication. Once this category is filled, only patients who are not on any preventative medications can be randomized into the study.

Major Exclusion Criteria:

* History of cluster headache.
* Presence of headaches more than 26 days a month on average for the 6 months prior to Screening.
* Failed to benefit from an adequate dose and duration, in the investigator's judgment (eg, one month of β-blocker), of 3 or more migraine preventive medications.
* Use of opiates or barbiturates more than 4 days per month for more than 3 consecutive months prior to Visit 1 and during the study.
* Use of over-the-counter (OTC) nasal products (ie, saline spray, Neti-Pot, Naväge® etc.) during the study.
* Any use of intranasal corticosteroid medications or conditions in which use of intranasal corticosteroids may be indicated during the study, eg, unstable allergic rhinitis that has previously required intranasal corticosteroids. Intranasal corticosteroid use is not allowed within 28 days of Baseline/Randomization/Visit 2 and during the treatment phase or follow-up period of the study.
* Patients who recently discontinued treatment with an anti-calcitonin-gene-related peptide (CGRP) or participated in anti-CGRP clinical study must be at least 4 months from the last drug administration prior to Visit 1.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Sullivan, MD, Study Director — Tonix Pharmaceuticals
Locations (26):
- United States (26):
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Synergy Research Centers - Synergy San Diego, Lemon Grove, California
  - Excell Research, Oceanside, California
  - Viking Clinical Research, LTD, Temecula, California
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Segal Trials - Miami Lakes Medical Research Outpatient Site, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Diamond Headache Clinic, Chicago, Illinois
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Alliance for Multispecialty Research - Wichita West, Wichita, Kansas
  - DelRicht Research - LCMC Health Urgent Care, New Orleans, Louisiana
  - DelRicht Research - Neighborhood Health, Prairieville, Louisiana
  - Boston Clinical Trials, Inc., Boston, Massachusetts
  - Michigan Headache & Neurological Institute, Ann Arbor, Michigan
  - DelRicht Research - Gulfport Memorial, Gulfport, Mississippi
  - Clinvest Research, Springfield, Missouri
  - Alliance for Multispecialty Research - Las Vegas, Las Vegas, Nevada
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - Peters Medical Research, High Point, North Carolina
  - IPS Research Company, INC., Oklahoma City, Oklahoma
  - DelRicht Research - Grassroots Healthcare, Tulsa, Oklahoma
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Austin Clinical Trial Partners, Austin, Texas
  - Charlottesville Medical Research, LLC, Charlottesville, Virginia
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Started | 27 | 31 | 30
Completed | 25 | 26 | 27
Not Completed | 2 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose | Total
Number analyzed (Participants) | 27 | 31 | 30 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (10.61) | 40.0 (10.93) | 44.1 (11.43) | 42.1 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 12
  Male | 21 | 27 | 28 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 2 | 12
  Not Hispanic or Latino | 21 | 27 | 28 | 76
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 6 | 6 | 14
  White | 24 | 22 | 22 | 68
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 27 | 31 | 30 | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Number of Monthly Migraine Headache Days
Description: Mean change in the number of monthly migraine headache days from the last 28 days of Baseline to the last 28 days of treatment (ie, month 3). A migraine headache day is any calendar day (0:00 to 23:59) in which the patient records in the e-diary:
  * An attack lasting 4 hours or more and meeting the ICHD-3 criteria for migraine without aura, or
  * A migraine with aura, or
  * An attack that meets ICHD-3 criteria for probable migraine, (a migraine subtype fulfilling all but one criteria (B-D) for migraine without aura), or
  * An attack of any duration that was believed by the patient to be a migraine and was relieved by a triptan, ergot derivative, or other migraine-specific abortive medication.
Time Frame: Last 28 days before Visit 2 (Day 1) and last 28 days before Visit 5 (Week 12)
Population: Data is reported for the mITT population, which includes all randomized patients who received at least one dose of study drug and had at least one post-Baseline evaluable month (that is, at least one of the three 28-day periods has at least 14 non-missing e-diary entries).
Measure: Least Squares Mean (Standard Error); unit: number of days
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
number of days | -8.17 (1.366) | -7.78 (1.246) | -5.77 (1.301)

2. Secondary Outcome: Proportion of Patients Experiencing a ≥ 50% Reduction in the Number of Migraine Headache Days
Description: Proportion of patients experiencing a ≥ 50% reduction in the number of migraine headache days from the last 28 days of Baseline to the last 28 days of treatment in each treatment group
Time Frame: Last 28 days before Visit 2 (Day 1) treatment and last 28 days before Visit 5 (Week 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
Participants | 15 | 15 | 10

3. Secondary Outcome: Mean Change in the Number of Days Using Rescue Medication
Description: Mean change in the number of days using rescue medication (triptan, ergot derivative, or other migraine-specific acute medication) from the last 28 days of Baseline to the last 28 days of treatment.
Time Frame: Last 28 days before Visit 2 (Day 1) treatment and last 28 days before Visit 5 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
days | -3.16 (.749) | -4.09 (.687) | -2.07 (.715)

4. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: Proportion of patients with a Patient Global Impression of Change (PGIC) of 1, "very much improved", or 2, "much improved", at Week 12. Scores range from 1 to 7. Lower scores indicate more improvement.
Time Frame: Visit 5 (Week 12)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
Participants | 12 | 16 | 14

5. Secondary Outcome: Mean Change in the Number of Moderate or Severe Headache Days
Description: Mean change in the number of moderate or severe headache days from the last 28 days of Baseline to the last 28 days of treatment. A moderate or severe headache day is defined as any calendar day wherein a patient records a headache or migraine of moderate or severe peak intensity in the e-diary.
Time Frame: Last 28 days before Visit 2 (Day 1) and last 28 days before Visit 5 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
days | -8.39 (1.372) | -8.17 (1.236) | -5.00 (1.304)

6. Secondary Outcome: Mean Change in the Number of Migraine Headache Days
Description: Mean change in the number of migraine headache days from the last 28 days of Baseline to average number per 28 days over the entire 12-week duration of Treatment Period.
Time Frame: Last 28 days before Visit 2 (Day 1) and average per 28 days over 12-week Treatment Period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
days | -7.09 (1.208) | -6.67 (1.063) | -5.24 (1.146)

7. Secondary Outcome: Mean Change From Baseline in the Migraine-Specific Quality of Life Questionnaire
Description: Mean change from Baseline in the Migraine-Specific Quality of Life Questionnaire (MSQ v2.1) at Week 12. Scores range from 0 to 100. Higher scores indicate better quality of life.
Time Frame: Visit 2 (Day 1) and Visit 5 (Week 12)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
Number analyzed (Participants) | 27 | 31 | 29
units on a scale | 26.07 (4.154) | 28.98 (3.727) | 21.10 (3.928)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | TNX-1900 Low Dose | TNX-1900 High Dose
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 6/27 | 10/31 | 5/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=27) | TNX-1900 Low Dose (N=31) | TNX-1900 High Dose (N=30)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 10 | 5
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Migraine (Nervous system disorders) | 0 | 2 | 0
Product after taste (Product Issues) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An industry standard NDA is in place with all investigators.

DOCUMENTS (2):
  • Study Protocol (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT05679908/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT05679908/SAP_001.pdf